CLINICAL TRIAL: NCT06017739
Title: Hypersecreting Patients (COPD And/or Bronchiectasic) Comparing 2 Technologies: Efa vs Efa + High Flow
Brief Title: Expiratory Flow Accelerator (Efa) vs Efa + High Flow in Chronic COPD and Bronchiectasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale della Valle Olona (Other)
Responsible Party: Principal Investigator, MARIANNA MESSINA, Principal Investigator, Azienda Socio Sanitaria Territoriale della Valle Olona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 759del07/08/23
Record Dates: First submitted 2023-08-18; First posted 2023-08-30 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Copd; Bronchiectasis Adult
Keywords: EFA; HIGH FLOW; BRONCHIECTASIS; COPD; HYPERSECRETION
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiectasis

STUDY DESIGN:
Intervention Model Description: the two arms of the study are:
  1. EFA / EFA + High Flow
  2. EFA + High Flow / EFA patients are randomly assigned to one of two groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expiratory Flow Accelerator (Experimental): Patients for 6 weeks use the Expiratory Flow Accelerator Technology
  Interventions: Device: Bronchial Clearance A
- Expiratory Flow Accelerator + HIGH FLOW Technology (Experimental): Patients for 6 weeks use the EFA technology and High Flow Technology
  Interventions: Device: Bronchial Clearance B

INTERVENTIONS:
Device: Bronchial Clearance A — EFA technology: the patient has to breathe at tidal volume by a mouthpiece at level 5 for half an hour twice a day.
  Arms: Expiratory Flow Accelerator
Device: Bronchial Clearance B — High Flow Technology: patient has to wear nasal cannula and breathe his nose for one hour twice a day. After he has to use EFA technology level 5 for half an hour twice a day.
  Arms: Expiratory Flow Accelerator + HIGH FLOW Technology

SUMMARY:
The aim of the study is to compare the efficacy of using EFA technology versus the combination of EFA + high flow in hypersecretory patients COPD and bronchiectasis

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a 13-weeks trial period: 6 weeks of one technology (EFA / EFA+ HIGH FLOW), 1- wash out week and 6- weeks of the other technology in a cross over randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosed by spirometry
* Bronchiectasis diagnosed by CT
* 2 Exacerbation/year

Exclusion Criteria:

* Cystic Fibrosis
* OSAS
* Non Invasive Ventilation
* Ineffective Cough
* Exacerbation in progress
* Hemodynamic Instability
* severe heart failure

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-07-18 (Estimated); Study Completion 2025-01-18 (Estimated)

PRIMARY OUTCOMES:
Cough Severity | "Day0", "Week6", Week13"
  Visual Analogic Scale (0=not severe cough;10=very severe cough)
Expectoration Difficulty | "Day0", "Week6", Week13"
  Visual Analogic Scale (0=not severe expectoration difficulty;10= very severe expectoration difficulty)

SECONDARY OUTCOMES:
FEV 1 (Forced Expiratory Volume) | "Day0", "Week6", Week13"
  Airway obstruction index measured by spirometry
Exacerbations | "Day0", "Week6", Week13"
  number of exacerbation/ year
Inspiratory Capacity | "Day0", "Week6", Week13"
  air trapping index measured by spirometry
6 minutes walking test | "Day0", "Week6", Week13"
  index of cardiorespiratory function in activities of daily living
Saint George Respiratory Questionnaire | "Day0", "Week6", Week13"
  quality of life
Medical Research Council mMRC | "Day0", "Week6", Week13"
  dyspnea perception (0 no dyspnea, 4 very important dyspnea)
SpO2 (Oxygen Saturation by Pulse Oximetry) | "Day0", "Week6", Week13"
  blood oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Messina, Principal Investigator — ASST Valle Olona
Locations (1):
- Marianna Messina, Somma Lombardo, Varese, Italy

IPD SHARING:
Plan to Share IPD: No